CLINICAL TRIAL: NCT00484458
Title: A Prospective, Multi-center, Randomized, Active-Controlled Study of the Wallis System for the Treatment of Mild to Moderate Degenerative Disc Disease of the Lumbar Spine
Brief Title: Wallis Stabilization System for Low Back Pain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zimmer Spine (Industry)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6000-1006-P1-R1
Record Dates: First submitted 2007-06-07; First posted 2007-06-11 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-10

CONDITIONS: Low Back Pain
Keywords: Degenerative Disc Disease; Total Disc Replacement
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Degeneration | interventions — Total Disc Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Wallis Stabilization System
  Interventions: Device: Interspinous process and dynamic stabilization (Wallis System)
- 2 (Active Comparator): Total Disc Replacement
  Interventions: Device: Total Disc Replacement

INTERVENTIONS:
Device: Interspinous process and dynamic stabilization (Wallis System) — Interspinous stabilization
  Arms: 1
Device: Total Disc Replacement — Total disc
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate that the Wallis System (interspinous process implant) is equivalent to total disc replacement (TDR) for the treatment of mild to moderate degenerative disc disease (DDD) of the lumbar spine at the L4-L5 level.

This study will assess the safety and efficacy of the Wallis® System compared to commercially available lumbar TDR with respect to individual subject success rates at 24 months postoperative follow-up.

Study participants will receive all study related test articles and surgical procedures at no charge. Please scroll down to the "Locations" section to find a doctor in your area that is participating in this study. If you are interested in participating in this study and do not see a doctor in your area, please contact Jose Naveira at jose.naveira@abbottspine.com

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 (inclusive) and skeletally mature.
* Diagnosis of mild to moderate DDD at L4-L5 as confirmed by radiography.
* Minimum of six months of failed conservative treatment.
* Pre-operative visual analog (VAS) low back pain score ≥ 40, on a scale of 100mm, with low back pain greater than left or right leg pain.
* Preoperative baseline Oswestry Disability Index (ODI) score of ≥ 40 on a 100 point scale.
* Physically and mentally able to comply with the protocol, including ability to read and complete required forms, and willing and able to adhere to the follow-up requirements of the protocol.
* Voluntarily signs the patient informed consent form.
* Patient is a surgical candidate for an anterior approach to the lumbar spine (< 3 abdominal surgeries).

Exclusion Criteria:

* The investigator believes that the L1-L2, L2-L3, L3-L4, or L5-S1 level is symptomatic based upon objective evidence, e.g., radiograph, MRI, or discography.
* Evidence of a prior fracture or trauma to the vertebral bodies at the affected level and/or the spinous processes at the L4-L5 or adjacent levels.
* Osteoporosis or osteopenia or metabolic bone disease as confirmed by DEXA scan (T score < -1.0). Female subjects older than 45 years of age (or post-menopausal women, history of oophorectomy, or family history of osteoporosis) and male subjects older than 55 years will undergo a pre-operative, dual energy x-ray absorptiometry (DEXA) of the lumbar spine. The DEXA will be used to identify subjects with an indication of osteoporosis, osteopenia or metabolic bone disease. Subjects with a T-score of less than -1.0 will be excluded from the study.
* Congenital lumbar spinal stenosis.
* Bony lumbar stenosis.
* Extreme obesity, as defined by National Institutes of Health (NIH) Clinical Guidelines Body Mass Index (BMI > 40kg/m2).
* A history of any surgical procedure intended to remove or alter the disc (e.g. discectomy, intradiscal electrothermal therapy (IDET) or enzymes), decompress (laminectomy) or fuse, either the index or adjacent levels.
* Prior participation in study of any investigational spinal implant or investigational spinal treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 340 (Estimated)
Dates: Start 2007-01; Primary Completion 2013-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Non-inferior to commercially available lumber TDR after 24 months. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: John J. Regan, MD, Principal Investigator — Spine Source; Christopher Bergin, MD, Principal Investigator — Illinois Bone & Joint Institute
Locations (11):
- United States (11):
  - Spine Source, Beverly Hills, California
  - Core Orthopaedic Medical Center, Encinitas, California
  - Boulder Neurosurgical Associates, Boulder, Colorado
  - Denver Spine, Greenwood Village, Colorado
  - Illinois Bone & Joint Institute, Morton Grove, Illinois
  - Fort Wayne Orthopaedics, Fort Wayne, Indiana
  - Medical University of South Carolina, Charleston, North Carolina
  - Triangle Orthopaedic Associates, P.A., Durham, North Carolina
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - University of Utah-Dept. of Neurosurgery-Dept. of Orthopedic Surgery, Salt Lake City, Utah
  - Aurora BayCare Medical Center, Green Bay, Wisconsin